CLINICAL TRIAL: NCT05606536
Title: The Impact of Intra-operative Fluid Infusion Rate on Hemodilution and Microcirculation Prospective Observational Pilot Study
Brief Title: The Impact of Intra-operative Fluid Infusion Rate on Microcirculation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Hradec Kralove (Other)
Responsible Party: Principal Investigator, David Astapenko, MD, PhD, Deputy Head for Science and Research, University Hospital Hradec Kralove
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CooperatioUK_MIC_HEM
Record Dates: First submitted 2022-10-26; First posted 2022-11-04 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Fluid Therapy; Microcirculation; Hemodilution
MeSH Terms: interventions — Crystalloid Solutions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- 10 % hemodilution (Experimental): Recumbent surgery:
  * infusion rate in first 20 minutes: 15 ml/kg/h
  * infusion rate after 20 minutes: 2,6 ml/kg/h
  Laparoscopic surgery:
  * infusion rate in first 20 minutes: 16 ml/kg/h
  * infusion rate after 20 minutes: 0,8 ml/kg/h
  Interventions: Drug: Crystalloid Solutions
- 20 % hemodilution (Experimental): Recumbent surgery:
  * infusion rate in first 20 minutes: 26 ml/kg/h
  * infusion rate after 20 minutes: 3,4 ml/kg/h
  Laparoscopic surgery:
  * infusion rate in first 20 minutes: 28 ml/kg/h
  * infusion rate after 20 minutes: 1,6 ml/kg/h
  Interventions: Drug: Crystalloid Solutions
- 30 % hemodilution (Experimental): Recumbent surgery:
  * infusion rate in first 20 minutes: 38 ml/kg/h
  * infusion rate after 20 minutes: 5,1 ml/kg/h
  Laparoscopic surgery:
  * infusion rate in first 20 minutes: 44 ml/kg/h
  * infusion rate after 20 minutes: 2,4 ml/kg/h
  Interventions: Drug: Crystalloid Solutions
- Standart care (No Intervention): Infusion rate based upon the standard care.

INTERVENTIONS:
Drug: Crystalloid Solutions — Locally approved crystalloid solution will be given at the predefined infusion rate
  Arms: 10 % hemodilution; 20 % hemodilution; 30 % hemodilution

SUMMARY:
Intraoperative fluid therapy (IFT) is an integral part of anesthesia care during surgery. Its main indication is the optimization of oxygen supply to the tissues. For elective surgery that is not associated with higher blood loss and a long period of preoperative fasting, including fluids IFT is dosed to cover the basal daily need for fluids. However, it is not clear whether this fluid dose is optimal. Surgery is a stress factor that leads, among other things, to damage of the endothelial glycocalyx (EG). EG binds a significant amount of plasma, which is released during EG destruction and causes relative hemodilution.

Isovolumic hemodilution is an established intraoperative procedure that serves to better control bleeding in procedures where bleeding is expected. However, partial hemodilution occurs even with standard IFT, and even when fluids are hardly given at all. Flow parameters in microcirculation have not yet been described depending on IFT conduction. The parameters of the microcirculation reflect its functioning, which will consequently affect the postoperative phase of the patient's moaning and clinical outcome.

DETAILED DESCRIPTION:
Intraoperative fluid therapy (IFT) is an integral part of anesthesia care during surgery. Its main indication is the optimization of oxygen supply to the tissues. IFT is tailored to the surgical performance, blood loss, and patient (comorbidities, length of preoperative fasting, hydration level, volemia status). For elective surgery that is not associated with higher blood loss (< 200 ml) and a long period of preoperative fasting, including fluids (fluids per os < 2 hours before the procedure), IFT is dosed to cover the basal daily need for fluids (approx. 1-2 ml) /kg.hour-1). However, it is not clear whether this fluid intake is optimal. Surgery is a stress factor that leads, among other things, to damage of the endothelial glycocalyx (EG), which is a thin carbohydrate layer on the endoluminal side of endothelial cells, which is of fundamental importance for the physiology of microcirculation and tissue metabolism. EG also binds a significant amount of plasma (estimated up to 1.7 liters), which is released during EG destruction and causes relative hemodilution.

Isovolumic hemodilution is an established intraoperative procedure that serves to better control bleeding in procedures where bleeding is expected (e.g. cardiac surgery using an extracorporeal circuit or vascular surgery). However, partial hemodilution occurs even with standard IFT, and even when fluids are hardly given at all. Flow parameters in microcirculation have not yet been described depending on IFT conduction. The parameters of the microcirculation reflect its functioning, which will consequently affect the postoperative phase of the patient's moaning and clinical outcome.

ELIGIBILITY:
Inclusion Criteria:

* elective recumbent and laparoscopic surgery
* informed consent

Exclusion Criteria:

* blood loss over 250 ml
* hemodynamic instability requiring noradrenaline infusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Sublingual microcirculation profile | 1 hour
  During one hour four measurements each 20 minutes will take place. Recordings will be assessed automatically by specialised software. Microcirculatory parameters of interest are:
  capillary density, De Backer score, perfused capillary density and proportion of perfused vessels.
  Capillary density comes in mm/mm2 and the higher number the better, there is not approved median number.
  De Backer score is derived from capillary density and it is without dimension. Perfused capillary density signifies a percent of perfused vessels and it is in %. Normal values in healthy adults are around 90 %.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Hradec Kralove, Hradec Králové, Czechia

IPD SHARING:
Plan to Share IPD: No